CLINICAL TRIAL: NCT07003711
Title: Effects of Progressive Muscle Relaxation Training Applied in Addition to Aerobic Exercise Training in Individuals With Migraine Diagnosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Hafize ALTAY, Principal Investigator, Mardin Artuklu University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/7-8
Record Dates: First submitted 2025-05-20; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Migraine Disease
Keywords: aerobic exercise; physical therapy; therapy; migraine; relaxation
MeSH Terms: conditions — Migraine Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants who meet the inclusion criteria will be randomly assigned to one of two groups: exercise or control group. The exercise group will be given both aerobic exercise and progressive muscle relaxation training. The control group will only receive aerobic exercise.
Who Masked: Outcomes Assessor
Masking Description: The evaluator will be blinded to the group assignments in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The exercise group will receive aerobic exercise and progressive muscle relaxation training.
  Interventions: Other: aerobic exercise and relaxation trainig
- Control Group (Active Comparator): The control group will receive aerobic exercise.
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise and relaxation trainig — Aerobic exercise and progressive muscle relaxation training will be given to the exercise group.
  Arms: Exercise Group
Other: aerobic exercise — Aerobic exercise will be applied to the control group.
  Arms: Control Group

SUMMARY:
Aim: The purpose of this study is to evaluate the effects of progressive muscle relaxation training, in addition to aerobic exercise training, on pain, disability, quality of life, psychological status, and functional capacity in individuals diagnosed with migraine.

Methods: The study population comprises migraine patients who presented to the Neurology Clinic of Mardin Training and Research Hospital. Participants meeting the inclusion criteria will be randomized into two groups: an exercise group and a control group. The exercise group will receive both aerobic exercise and progressive muscle relaxation training, while the control group will receive only aerobic exercise. Participants' physical and demographic characteristics, as well as migraine-associated symptoms, will be assessed and recorded. Pain characteristics will be evaluated using a pain diary and pressure pain threshold measurements of the head and neck muscles. Disability will be assessed with the Migraine Disability Assessment Scale (MIDAS). Quality of life will be measured using the Headache Impact Test (HIT-6). Psychological status will be evaluated with the Hospital Anxiety and Depression Scale (HADS). Functional capacity will be assessed clinically using the 6-Minute Walk Test.

DETAILED DESCRIPTION:
Participants in both groups will receive sessions under the supervision of a physiotherapist, three sessions per week for 12 weeks. The aerobic exercise program will consist of a warm-up, a main exercise phase (loading program), and a cool-down period. Progressive muscle relaxation training will be implemented as part of the relaxation training protocol.

ELIGIBILITY:
The inclusion criteria are listed as follows:

* Having been diagnosed with migraine by a specialist neurologist.
* Experiencing at least 3 migraine attacks per month.
* Being between the ages of 18 and 65.
* Volunteering to participate in the study.

Exclusion Criteria listed as follows:

* Being pregnant.
* Having any neurological disease other than migraine.
* Having other secondary headaches in addition to migraine.
* Having a recent history of head or neck trauma.
* Participating in a regular exercise program in the last 6 months.
* Having a history of malignancy.
* Having a disease or disability that may prevent aerobic exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Migraine-Related Disability Status Questionnaire | 12 week (before and after treatment)
  The Migraine Disability Assessment Scale (MİDAS) will be used to determine the level of inadequacies in daily activities of individuals with migraine. MIDAS is a scale that aims to evaluate the disability status related to headache and the functionality of individuals with migraine in daily and social activities. The MIDAS scale includes 5 questions regarding workplace, school, home work and social relationships.
Headache Impact Questionnaire (HIT-6) | 12 weeks (before and after treatment)
  The Headache Impact Questionnaire (HIT-6) will be used to assess the quality of life due to headache in individuals with migraine. The Turkish validity and reliability of the scale was performed by Dikmen and colleagues. It consists of 6 questions including the frequency of headache, the ability to carry out daily activities due to headache, the degree of limitation in social life, the need for rest, and the change in mood. This scale can be scored between 36 and 78. Higher scores on this scale indicate that the individual's quality of life is affected.
Hospital Anxiety and Depression Scale | 12 weeks (before and after treatment)
  Hospital Anxiety and Depression Scale (HADS) is a self-report scale developed to determine the risk of anxiety and depression and to measure the level and severity of change. The Turkish version of the scale was found to be valid and reliable. HADS is a 14-item self-assessment scale used to evaluate anxiety and depression levels. It consists of two subscales-7 items each for anxiety (HADS-A) and depression (HADS-D), scored from 0 to 21 (0-7 normal, 8-10 mild, 11-14 moderate, 15-21 severe). Higher scores indicate higher levels of anxiety or depression.
6 min Walking Test | 12 weeks (before and after treatment)
  The 6-minute walk test is used as a simple measure of aerobic exercise capacity. The test involves walking on a flat surface for 6 minutes according to a standardized protocol. The distance walked before and after the 6-minute test will be recorded in meters.
pain diary | 20 weeks (4 weeks before treatment, 12 weeks during treatment, 4 weeks after treatment)
  Pain diaries are considered the gold standard for individuals with headaches. The severity of headaches during attacks, their duration (minutes), frequency, possible triggering factors, and the amount and type of medication taken will be recorded. The average pain intensity during headache attacks experienced by individuals with migraine in the last month will be assessed using the Numerical Pain Rating Scale (NADS), which has a score between 0 and 10 .
pressure pain threshold assessment | 12 weeks (before and after treatment)
  The pressure algometer is recognized as an objective method for assessing pain threshold. A pressure of approximately 1 kg/cm² will be applied to designated motor points of the muscles using the disk head of the algometer device, positioned at a 90-degree angle perpendicular to the skin. Participants will be instructed to say "stop" at the moment they first perceive pain. To ensure participant adaptation prior to the actual test, three consecutive measurements will be conducted for each muscle, with a 1-minute interval between measurements, and the average score will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda TOPRAK ÇELENAY, professor, Study Director — Ankara Yildirim Beyazıt University

IPD SHARING:
Plan to Share IPD: No
Study data cannot be shared as it will contain personal information.